CLINICAL TRIAL: NCT02551146
Title: Influence of Implants and Locators for Improved Retention of Mandibular Full Dentures on Patient's Quality of Life and Oral Function. A Controlled, Randomized and Prospective Study
Brief Title: Influence of Implants and Locators for Improved Retention
Acronym: GC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties concerning the recruitment of participants
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKS-217
Record Dates: First submitted 2015-09-03; First posted 2015-09-16 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Locator with retention elements (Experimental): GC Pilier Locator abutment with retention elements:
  For patients in the experimental group (arm A) the connection of the full dentures to the implants will be achieved by fitting the dentures with GC Pilier Locator abutments with retention elements.
  Interventions: Device: A Locator with retention elements
- B Locator without retention elements (Active Comparator): GC Pilier Locator abutment without retention elements:
  For patients with the active comparator (arm B) the full dentures will get Pilier Locator abutments without retention elements and thus no connection to the implants.
  Interventions: Device: B Locator without retention elements

INTERVENTIONS:
Device: A Locator with retention elements — Insertion of GC Pilier locator abutments with retention elements
  Arms: A Locator with retention elements
Device: B Locator without retention elements — Insertion of GC Pilier locator abutments without retention elements
  Arms: B Locator without retention elements

SUMMARY:
The aim of this study is to assess the influence of this particular treatment method on the patients' quality of life and masticatory function.

DETAILED DESCRIPTION:
For this prospective randomized controlled clinical trial patients with edentulous mandibles and tissue supported (full) dentures were treated with 2 dental implants and locators in order to improve prosthesis stability.

The LOCATOR System is comprised of three parts: The LOCATOR implant attachment (LOCATOR abutment), the LOCATOR Male and the LOCATOR Denture Cap. The abutment is inserted directly into the implant using a torque wrench, while the Denture Cap is placed into the base of the overdenture for polymerization using acrylic resin. Custom retention is achieved via LOCATOR Males - small color-coded (according to retention force) plastic inserts - which can be exchanged as needed.

ELIGIBILITY:
Inclusion Criteria:

* age 45-80 years (male or female)
* sufficient full dentures in the mandible
* must be able to clean their teeth on their own
* edentulous mandible with interforaminal adequate bone for insertion of implants
* implantation sites free of infections and root fragments
* no need for treatment of the maxillary teeth
* Written Informed Consent

Exclusion Criteria:

* systemic diseases
* mental disability that may affect the participant's ability to properly follow study instructions
* oral mucosal diseases
* long-term medication with steroids, bisphosphonates
* known allergic reactions to dental materials
* malignant tumor in the head and neck area
* requirement of any concurrent radiotherapy or chemotherapy or any radiotherapy or chemotherapy within the last 10 years pregnancy or breastfeeding at study entry

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Quality of life (OHIP-G-49) | 3 months after randomization
  The oral health-related quality of life is assessed by the German version of the Oral Health Impact Profile questionnaire (OHIP-G-49, Locker et al 1993)

SECONDARY OUTCOMES:
masticatory function | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  Video documentation of chewing a defined bolus. After chewing a defined bolus for 10 seconds comparison of reduction ratio of the bolus is documented by photography and the change from baseline will be documented.
Plaque index | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The Plaque index (Silness and Loe 1964) will be assessed and the change from baseline will be documented.
Probing pocket depth | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The Probing pocket depth with bleeding on probing (6 sites of every tooth and implant) will be assessed and the change from baseline will be documented.
Gingival index | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The Gingival index (Loe and Silness 1963) will be assessed and the change from baseline will be documented.
Gingival recessions | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The Gingival recessions at teeth will be assessed and the change from baseline will be documented.
Mucosal recessions | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The mucosal recessions at implants will be assessed and the change from baseline will be documented.
width of keratinized gingiva/mucosa | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  The width of keratinized gingiva/mucosa will be assessed and the change from baseline will be documented.
intraoral photo-documentation | 3 months (T0), 6 months (T1), 9 months (T2), 12 months (T3)
  A photo-documentation (intraoral) will be done to assess the changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Reiner Mengel, Professor MD, Principal Investigator — Dept. of Prosthodontics and Orofacial Function Philipps-University, School of Dental Medicine
Locations (1):
- Dept. of Prosthodontics and Orofacial Function Philipps-University, School of Dental Medicine, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assuncao WG, Barao VA, Delben JA, Gomes EA, Tabata LF. A comparison of patient satisfaction between treatment with conventional complete dentures and overdentures in the elderly: a literature review. Gerodontology. 2010 Jun;27(2):154-62. doi: 10.1111/j.1741-2358.2009.00299.x. Epub 2009 May 6. PMID 19467020